CLINICAL TRIAL: NCT01113346
Title: Phase II Double Blind Placebo-controled Randomized Comparative Multicentered Study of Efficacy and Safety of Filtrum-STI, 0,4g Tablets (Produced by AVVA RUS) in Children With Viral Gastroenteritis
Brief Title: A Pilot Study of Filtrum-STI in Children With Viral Gastroenteritis
Acronym: F-GE-09
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Avva Rus, JSC (Industry)
Collaborators: St. Vladimir Moscow Children's Clinical Hospital (Unknown); Arhangelsk Regional Children's Clinical Hospital named after Vizshletsov P.G. (Unknown)
Responsible Party: Dr. Elena Meskina, MD, DrSc, St. Vladimir Moscow Children's Clinical Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 03/09-AVVA RUS
Record Dates: First submitted 2010-04-12; First posted 2010-04-29 (Estimated); Last update posted 2010-07-14 (Estimated); Status verified 2010-07

CONDITIONS: Viral Gastroenteritis
Keywords: enterosorbent; sorbent; gastrointestinal decontamination; viral diarrhea; rotavirus; Filtrum; Filtrum-STI; lignin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Filtrum-STI (Experimental)
  Interventions: Drug: Filtrum-STI (lignin hydrolytic)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Filtrum-STI (lignin hydrolytic) — For children aged less than 1 y.o.: Filtrum-STI, 400mg per day (1/2 tablet 2 times a day) for 7 days.
  For children aged 1-4 y.o.: Filtrum-STI, 800mg per day (1 tablet 2 times a day) for 7 days.
  Other Names: lignin hydrolytic, sorbent, enterosorbent
  Arms: Filtrum-STI
Drug: Placebo — For children aged less than 1 y.o.: Placebo, 1/2 tablet 2 times a day for 7 days.
  For children aged 1-4 y.o.: Placebo, 1 tablet 2 times a day for 7 days.
  Arms: Placebo

SUMMARY:
This is a phase II double blind multicenter randomized placebo-controled clinical study aimed to find out whether treatment with Filtrum-STI (orally administered 0,4g tablets) is safe and effective in children with viral gastroenteritis. Filtrum-STI (lignin hydrolytic) is a drug with a high absorbing ability, that binds and eliminates toxins, pathogenic microorganisms and viruses. Filtrum-STI is inoffensive for mucous membranes, enhances colonic propulsion and improves its natural microflora. The drug is not toxic and well combines with other medication

ELIGIBILITY:
Inclusion Criteria:

* children aged 0-4 y.o. diagnosed with moderate viral gastroenteritis;
* 72 h or less from the onset of gastrointestinal symptoms.

Exclusion Criteria:

* severe diseases;
* individual intolerance of Filtrum-STI
* treatment with antiviral, immunomodulatory drugs during the study and 2 weeks before inclusion
* treatment with pre- pro- and antibiotics 2 weeks before inclusion
* participation in other clinical study 1 month before inclusion and during participation in the study.

Ages: 1 Month to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-12 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Severity of gastroenteritis | Day 7 after start of the intervention
  It's measured by ordinal scales (4- and 5-scores) using data about patients' body temperature, bloating, nausea, abdominal pain, meteorism, stool frequency (physical examination and parent-reported questionnaire).

SECONDARY OUTCOMES:
Intestinal Viruses detection and quantification | Day 7 after start of the intervention
  It is measured by PCR laboratory test
Secretory IgA | Day 7 after start of the intervention
Severity of gastroenteritis | Day 10-14 after end of the intervention
  It's measured by ordinal scales (4- and 5-scores) using data about patients' body temperature, bloating, nausea, abdominal pain, meteorism, stool frequency (physical examination and parent-reported questionnaire).
Scatological examination | Day 7 after start of the intervention
Scatological examination | Day 10-14 after end of the intervention
Dysbacteriosis analysis | Day 7 after start of the intervention
Intestinal Viruses detection and quantification | Day 10-14 after end of the intervention
Secretory IgA | Day 10-14 after end of the intervention
Vital functions | Days 1,2,3,4,5,6,7 after start of the intervention and day 10-14 after end of one
  It includes Heart rate, Breathing rate, Body temperature.
Blood test | Day 7 after start of the intervention
Biochemical blood analysis | Day 7 after start of the intervention
  It includes crude protein, alanine aminotransferase, aspartate aminotransferase, bilirubin, blood urea, creatinine, sodium, potassium, glucose.
Urine analysis | Day 7 after start of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Elena Meskina, MD, DrSc, Principal Investigator — St. Vladimir Children's Moscow Clinical Hospital; Lyudmila Kobeleva, MD, PhD, Study Director — Avva Rus, JSC; Nickolay A. Kryuchkov, MD, PhD, MPH, Study Director — Avva Rus, JSC
Locations (2):
- Russia (2):
  - Arhangelsk Regional Children's Clinical Hospital named after P.G. Vizshletsov, Arhangelsk, Arhangelskaya Oblast
  - St. Vladimir Children's Moscow Clinical Hospital, Moscow, Moscow